CLINICAL TRIAL: NCT01779401
Title: Investigator Initiated Prospective Study to Investigate the Best Anti-platelet Treatment in High Thrombotic Risk PCI Patients.
Brief Title: Clopidogrel Response Evaluation and AnTi-Platelet InterVEntion in High Thrombotic Risk PCI Patients
Acronym: CREATIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Beijing Municipal Health Bureau (Other); Haemonetics Corporation (Industry); Zhejiang Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yi-Da Tang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-4003-03
Record Dates: First submitted 2013-01-15; First posted 2013-01-30 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Coronary Heart Disease
Keywords: PCI; platelet function monitoring; Thrombelastography; clopidogrel; cilostazol; in-stent thrombosis
MeSH Terms: conditions — Coronary Disease | interventions — Clopidogrel; Aspirin; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clopidogrel + Aspirit (Active Comparator): A Standard antiplatelet therapy control group： Clopidogrel 75mg Qd + Aspirin 100mg Qd
  Interventions: Drug: Clopidogrel 75mg; Drug: Aspirin 100mg
- Clopidogrel + Aspirin (Active Comparator): B Double-dosage Clopidogrel group： Clopidogrel 150mg Qd + Aspirin 100mg Qd
  Interventions: Drug: Clopidogrel 150mg; Drug: Aspirin 100mg
- Clopidogrel + Aspirin + Cilostazol (Active Comparator): C triple antiplatelet therapy group： Cilostazol 100mg Bid + Aspirin 100mg Qd + Clopidogrel 75mg Qd
  Interventions: Drug: Clopidogrel 75mg; Drug: Aspirin 100mg; Drug: Cilostazol 100mg

INTERVENTIONS:
Drug: Clopidogrel 75mg
  Arms: Clopidogrel + Aspirin + Cilostazol; Clopidogrel + Aspirit
Drug: Clopidogrel 150mg
  Arms: Clopidogrel + Aspirin
Drug: Aspirin 100mg
Drug: Cilostazol 100mg
  Arms: Clopidogrel + Aspirin + Cilostazol

SUMMARY:
To identify the high-risk patients who might have in-stent thrombosis after PCI with thromboelastography and to head-to-head compare two intensified antiplatelet therapeutic strategies of double-dosage Clopidogrel and triple antiplatelet therapy with Cilostazol with the standard antiplatelet therapy.

DETAILED DESCRIPTION:
Study population: Age 18 - 75, male or non-pregnant female; stable or unstable angina with evidence of myocardial ischemia, or patient with myocardial infarction; coronary angiography reveals stenosis lesions; discovery of ADP induced platelet inhibition rate < 50% and MAADP > 47mm via thromboelastography (indicating low responsiveness to Clopidogrel with high risk for stent thrombosis formation); is able to understand the objective of the trial, takes part voluntarily and signs the written informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75, male or non-pregnant female;
2. Stable or unstable angina with evidence of myocardial ischemia, or patient with myocardial infarction;
3. Coronary angiography reveals stenosis lesions;
4. Discovery of ADP induced platelet inhibition rate < 50% and MAADP >47mm via thromboelastography (indicating low responsiveness to Clopidogrel with high risk for stent thrombosis formation);
5. Is able to understand the objective of the trial, takes part voluntarily and signs the written informed consent form.

Exclusion Criteria:

1. Those who have participated in other drug or therapy equipment clinical trials but did not reach the main study endpoint time limit;
2. Symptoms of severe heart failure (NYHA Class III and above) or left ventricular ejection fraction < 40% (ultrasound or left ventricle ngiography);
3. Pregnant or lactating women;
4. severely impaired renal function before surgery: serum creatinine > 2.0mg/dl;
5. Impaired liver function before surgery: Serum GPT > 120U/L;
6. Bleeding tendency, history of active peptic ulcer, history of cerebral hemorrhage or cavum subarachnoidale bleeding, patients with antiplatelet agent and anticoagulant treatment contraindications and hence are unable to undergo anticoagulant therapy;
7. Patients who are unable to withstand dual antiplatelet therapy due to allergy to Aspirin, Clopidogrel or ticlopidine, heparin, contrast agent, paclitaxel and metals;
8. Leucocyte < 3.5 x 109; and/or platelet < 100,000/mm3 or > 750,000/mm3;
9. Patient's life expectancy is less than 12 months;
10. Patients who plan to undergo coronary artery bypass grafting or other surgery within 1 year;
11. Those waiting for heart transplant;
12. Patients who are deemed by the researchers to have low compliance and unable to abide by the requirements and complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1078 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | within 1.5years of patient enrolled
  MACCE, including cardiac death, myocardial infarction, target vessel revascularization and cerebrovascular events

SECONDARY OUTCOMES:
Secondary endpoint | within 1.5 years of patients enrolled
  Occurrence of stent thrombosis
bleeding | within 1.5 years of patients' enrolled
  Major bleeding and minor bleeding
quality of life of patient | within 1.5 years of patients' enrolled
  to evaluate with Seattle Angina Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, PHD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Cardiovascular Hospital, Beijing, China

REFERENCES:
- [Derived] Tang YD, Wang W, Yang M, Zhang K, Chen J, Qiao S, Yan H, Wu Y, Huang X, Xu B, Gao R, Yang Y; CREATIVE Investigators. Randomized Comparisons of Double-Dose Clopidogrel or Adjunctive Cilostazol Versus Standard Dual Antiplatelet in Patients With High Posttreatment Platelet Reactivity: Results of the CREATIVE Trial. Circulation. 2018 May 22;137(21):2231-2245. doi: 10.1161/CIRCULATIONAHA.117.030190. Epub 2018 Feb 2. PMID 29420189